CLINICAL TRIAL: NCT03794414
Title: The Influence of Positive End-expiratory Pressure (PEEP) in Predicting Fluid Responsiveness in Patients Undergoing One-lung Ventilation
Brief Title: Positive End-expiratory Pressure (PEEP) in Predicting Fluid Responsiveness in Patients Undergoing One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Choi Eun MI, Professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-11-028
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer; Lung Diseases
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fluid responder (Experimental): patients with 10% or more increase in stroke volume after fluid challenge. Both arms receive PEEP challenge.
  Interventions: Procedure: PEEP challenge
- fluid non-responder (Experimental): patients with no increase or less than 10% increase in stroke volume after fluid challenge. Both arms receive PEEP challenge
  Interventions: Procedure: PEEP challenge

INTERVENTIONS:
Procedure: PEEP challenge — apply PEEP 10 mmHg in one-lung ventilating patients.

SUMMARY:
The present study is to evaluate the effect of positive end-expiratory pressure (PEEP) in predicting fluid responsiveness in patients undergoing one-lung ventilation.

DETAILED DESCRIPTION:
Appropriate fluid challenge is crucial during lung surgery under one-lung ventilation. Applying PEEP in mechanically ventilating patients changes dynamic hemodynamic parameters (stroke volume variation, pulse pressure variation), which is more pronounced in hypovolemic patients. The aim of the present study is to evaluate the mechanically ventilating patients under one-lung ventilation requiring fluid resuscitation by applying PEEP to predict fluid responsiveness.

The investigators hypothesized that applying PEEP in one-lung ventilating patients can also change dynamic parameters and the magnitude of the change of stroke volume variation, pulse pressure variation can predict fluid responsiveness. The investigator applied PEEP 10 mmHg in one-lung ventilating patients and observed the dynamic parameters including stroke volume variation, pulse pressure variation and then infused 6ml/kg of crystalloid for fluid challenge and diagnosed fluid responsiveness as 10% increase of stroke volume after fluid challenge.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing lung surgery under one-lung ventilation

Exclusion Criteria:

* arrhythmia
* moderate to severe valvular heart disease moderate to severe pericardial effusion left ventricular ejection fraction < 40%
* moderate to severe chronic obstructive lung disease
* unable to insert oesophageal Doppler Monitor (ODM) probe ( esophageal stent, esophageal cancer, previous esophageal surgery, esophageal stricture, esophageal varices, pharyngeal pouch and severe coagulopathy )
* patient refusal
* cannot understand the protocol
* less than 50kg or over 100kg in weight

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
pulse pressure variation | 5 minutes after PEEP challenge
  Temporary increase of PEEP will be able to predict fluid responsiveness using increase of pulse pressure variation over 1%.

SECONDARY OUTCOMES:
stroke volume variation | 5 minutes after PEEP challenge
  Temporary increase of PEEP will be able to predict fluid responsiveness using increase of stroke volume variation over 1%.

CONTACTS AND LOCATIONS:
Overall Officials: Eun-mi Choi, Professor, Study Chair — Kangnam Sungshim Hospital
Locations (1):
- Kangnam Sungshim Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
However, I can always share if required.